CLINICAL TRIAL: NCT01770587
Title: A Sleep-Oriented Intervention for Suicidal Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Ann Bernert, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22393; K23MH093490 (NIH)
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Insomnia; Suicidal Ideation
Keywords: Insomnia; Sleep; Behavioral Medicine; Suicide; Suicidal Ideation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Suicidal Ideation; Suicide

ARMS (1):
- Behavioral Insomnia Treatment (Experimental): Brief Behavioral Insomnia Treatment
  Interventions: Behavioral: Behavioral Insomnia Treatment

INTERVENTIONS:
Behavioral: Behavioral Insomnia Treatment

SUMMARY:
An open-label trial to investigate the use of a behavioral insomnia treatment for suicidal ideation.

ELIGIBILITY:
* Age 18 or older
* Clinically significant sleep disturbances
* Diagnosis of depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation | Change from Baseline in Suicidal Ideation at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Bernert, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Dept. of Psychiatry and Behavioral Sciences, Stanford, California, United States